CLINICAL TRIAL: NCT03096366
Title: Does Blood Flow Restriction Training Improve Quadriceps Function After Arthroscopic Knee Surgery? A Randomized Clinical Trial
Brief Title: Does Blood Flow Restriction Training Improve Quadriceps Function After Arthroscopic Knee Surgery?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: Principal Investigator, Walter R Lowe, Professor and Chair, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-1047
Record Dates: First submitted 2017-03-23; First posted 2017-03-30 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Quadriceps Atrophy; ACL Reconstruction
Keywords: anterior cruciate ligament reconstruction
MeSH Terms: interventions — Blood Flow Restriction Therapy; Physical Therapy Modalities

STUDY DESIGN:
Masking Description: Blinding is not possible given the nature of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Physical therapy (PT) plus blood flow restriction (BFR) (Experimental): Physical therapy consists of two or three 90-minute sessions per week for 6 weeks and a minimum of 18 visits required for study inclusion. With BFR, exercises will be performed at 30% one-rep max with the BFR cuff placed around the proximal thigh and inflated to 80% of limb occlusion pressure (avg: 150 mmHg).
  Interventions: Device: Blood flow restriction; Other: Physical therapy
- Physical therapy (Active Comparator): Physical therapy consists of two or three 90-minute sessions per week for 6 weeks and a minimum of 18 visits required for study inclusion.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Device: Blood flow restriction — With BFR, exercises will be performed at 30% one-rep max with the BFR cuff placed around the proximal thigh and inflated to 80% of limb occlusion pressure (avg: 150 mmHg).
  Arms: Physical therapy (PT) plus blood flow restriction (BFR)
Other: Physical therapy — Physical therapy consists of two or three 90-minute sessions per week for 6 weeks and a minimum of 18 visits required for study inclusion.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of physical therapy (PT) plus BFR training compared to PT alone (without BFR training) after ACL reconstruction in patients who require extended limited weight bearing through assessment of patient reported outcomes and functional testing. The hypothesis is that PT plus BFR training will mitigate the loss of quadriceps muscle cross-sectional area, strength, and function while also improving early clinical and functional results.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament (ACL) reconstruction with concomitant meniscus or cartilage restoration procedures
* Adherence to modified weight bearing status before initiation of PT
* Expected participation in recreational or competitive sports after release to full activities

Exclusion Criteria:

* Unable to attend (or participate in) physical therapy
* Pregnancy
* Malignancy
* Fracture
* Peripheral vascular disease
* History of deep vein thrombosis (DVT)

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Quadriceps Muscle Cross-Sectional Area (CSA) as Assessed by Ultrasound | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery
Change in Quadriceps Muscle Cross-Sectional Area (CSA) as Assessed by Ultrasound | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery
Change in Quadriceps Muscle Cross-Sectional Area (CSA) as Assessed by Ultrasound | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery

SECONDARY OUTCOMES:
Change in Passive Range of Motion as Assessed by Goniometer | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery
Change in Passive Range of Motion as Assessed by Goniometer | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery
Change in Passive Range of Motion as Assessed by Goniometer | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery
Change in Active Range of Motion as Assessed by the Straight-Leg-Raise Test | at start of PT, 1 month after start of PT
  The uninvolved knee is bent 90 degrees as determined by a standard goniometer. The patient/participant is asked to raise the involved limb to the height of the tibial tuberosity of the uninvolved limb. Initiation of PT is 1 month after surgery.
Change in Active Range of Motion as Assessed by the Straight-Leg-Raise Test | at start of PT, 2 months after start of PT
  The uninvolved knee is bent 90 degrees as determined by a standard goniometer. The patient/participant is asked to raise the involved limb to the height of the tibial tuberosity of the uninvolved limb.Initiation of PT is 1 month after surgery.
Change in Active Range of Motion as Assessed by the Straight-Leg-Raise Test | at start of PT, 5 months after start of PT
  The uninvolved knee is bent 90 degrees as determined by a standard goniometer. The patient/participant is asked to raise the involved limb to the height of the tibial tuberosity of the uninvolved limb.Initiation of PT is 1 month after surgery.
Isometric quadriceps strength as Assessed by Dynamometer | 1 month after start of PT
  Initiation of PT is 1 month after surgery.
Isometric quadriceps strength as Assessed by Dynamometer | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Isokinetic quadriceps strength as Assessed by Dynamometer | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Thigh circumference (proximal, mid, distal) as Assessed by Measuring tape | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery.
Change in Thigh circumference (proximal, mid, distal) as Assessed by Measuring tape | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Thigh circumference (proximal, mid, distal) as Assessed by Measuring tape | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Balance Error Scoring System | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Balance Error Scoring System | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Overhead Squat Test | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Overhead Squat Test | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Y-Balance Test | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Y-Balance Test | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Single-Leg Squat Assessment | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Single-Leg Squat Assessment | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Vail Sport Test | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Vail Sport Test | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Landing Error Scoring System | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Landing Error Scoring System | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Single leg Hop Testing | 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Functional Performance as Assessed by Single leg Hop Testing | 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Activity as Assessed by Patient-Reported Score on the Marx Scale | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery.
Change in Activity as Assessed by Patient-Reported Score on the Marx Scale | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Activity as Assessed by Patient-Reported Score on the Marx Scale | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Activity as Assessed by Patient-Reported Score on the Tegner Activity Scale | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery.
Change in Activity as Assessed by Patient-Reported Score on the Tegner Activity Scale | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Activity as Assessed by Patient-Reported Score on the Tegner Activity Scale | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Knee Function as Assessed by Patient-Reported Score on the 2000 IKDC Subjective Knee Evaluation Form | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery.
Change in Knee Function as Assessed by Patient-Reported Score on the 2000 IKDC Subjective Knee Evaluation Form | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Knee Function as Assessed by Patient-Reported Score on the 2000 IKDC Subjective Knee Evaluation Form | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Kinesiophobia as Assessed by Patient-Reported Score on the Tampa Scale for Kinesiophobia | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery.
Kinesiophobia as Assessed by Patient-Reported Score on the Tampa Scale for Kinesiophobia | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Kinesiophobia as Assessed by Patient-Reported Score on the Tampa Scale for Kinesiophobia | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Physiological Impact of Returning to Sport After ACL Reconstruction Surgery as Assessed by Patient-Reported Score on the Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) Scale | at start of PT, 1 month after start of PT
  Initiation of PT is 1 month after surgery.
Change in Physiological Impact of Returning to Sport After ACL Reconstruction Surgery as Assessed by Patient-Reported Score on the Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) Scale | at start of PT, 2 months after start of PT
  Initiation of PT is 1 month after surgery.
Change in Physiological Impact of Returning to Sport After ACL Reconstruction Surgery as Assessed by Patient-Reported Score on the Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) Scale | at start of PT, 5 months after start of PT
  Initiation of PT is 1 month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Walter R Lowe, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States